CLINICAL TRIAL: NCT04107545
Title: Metabolic, Functional and Nutritional Responses to Weight Cycling in Athletes: The WAVE Study
Acronym: WAVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Laboratoire AME2P (Unknown); Université de Fribourg, Department of Endocrinology, Metabolism and Cardiovascular System (Unknown); University of Leeds, Appetite Control and Energy Balance Research (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RBHP 2019 DUCLOS; 2019-A00699-48 (Other: 2019-A00699-48)
Record Dates: First submitted 2019-09-20; First posted 2019-09-27 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Athletes
Keywords: weight cycling; sport; appetite; energy metabolism
MeSH Terms: conditions — Weight Cycling | interventions — Cardiomegaly, Exercise-Induced

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- athletes (Experimental): 48 elite athletes, 24 men and 24 women, experiencing regular weight cycling.
  Interventions: Behavioral: athletes

INTERVENTIONS:
Behavioral: athletes — Control of body temperature using the bodyCap temperature monitor that records body temperature for up to 48h (three times)

SUMMARY:
Many elite athletes are submitted to frequent rapid weight loss periods to meet their competition weight category and then experience weight cycling (lowing and gaining weight regularly). This weight cycling induce severe temporary energetic and metabolic changes and when repeated over time can lead to permanent metabolic adaptations that might favor metabolic disorders, body weight gain and body composition changes (favoring fat mass). The exact effects of this weight cycling are not clear yet, especially in terms of metabolic, energetics, nutritional functional and psychological impacts. Better understand these adaptations and their variations during weight loss and weight gain in regular weight cycler is of main importance to prevent these athletes for future health issues.

The aim of the present project if to assess these metabolic, functional, energetic and nutritional adaptations during weight loss, weight stable and weight gain periods in athletes experiencing regular weight cycling.

DETAILED DESCRIPTION:
After an inclusion visit to ensure the eligibility of athletes to complete the entire study, each subject will perform 3 experimental sessions of 2 visits each : i) two visits during a period of maintenance of body weight (CON); ii) two visits during weight loss (WL); iii) two visits during a weight regain (WG). The order of the periods (maintenance, loss or weight gain) will depend on the dynamics of the weight variations of each athlete (endurance sport and weight class) during the season and will therefore be individualized.

All experiments will be conducted in the same way for the CON, WL or WG session.

Upon arrival, each subject will perform a resting metabolism with continuous measurement of heart rate variability (≈ 30 min). Then, from 8:30, blood and saliva samples will be taken (≈ 10 min). Then (≈ 8:45), they will perform anthropometric and body composition measurements (waist circumference, hip circumference, bioimpedance, DXA) (≈ 30 min). Following these measurements (≈ 9:15), the subjects will eat a standardized breakfast and the report to food will be evaluated thanks to the Leeds Foods Preference Questionnaire before and after the meal. They will then be asked (≈ 10h) to complete the Profile of Mood State Questionnaire to measure the athlete's psychological state. Participants will then perform a measurement of muscle function (≈ 10:30).

During the second visit, carried out between 1 and 5 days after the first visit, the maximum aerobic capacity of the athletes will be evaluated by mid-morning stress test.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 18 to 35 (inclusive),
* exercising at least 4 sessions of endurance or weight-based sporting activities per week for a performance objective,
* having variations of at least 5% of their weight body during the last 3 sporting seasons (a sporting season corresponds to a year during which alternates the periods of training, recovery and participation in official competitions).
* Subject capable of providing informed consent to participate
* Subject with a social security insurance.

Exclusion Criteria:

* Medical or surgical history deemed by the investigator to be incompatible with the study.
* Presence of chronic pathology.
* Disorders of eating behavior.
* Subjects born very prematurely defined as a pregnancy inferior to 28 weeks.
* Subjects having used a treatment for a small stature (eg growth hormone).
* For women: irregular menstruation (changes in menstrual cycles ≥ 6 days).
* Sports subjects with a stable weight during the last three sporting seasons (weight variation <5%).
* Take medication that can change body temperature.
* Pregnant or lactating women.
* Subjects with gastrointestinal complications and / or contraindications to ingestion of the capsule (eg diverticulosis, inflammatory bowel disease, gastrointestinal surgery ...).
* Subjects needing MRI during ingestion of the capsule or having a pacemaker or other implanted electro-medical device.
* Person under guardianship or not subject to a social security scheme.
* Refusal to sign the information and consent leaflet.
* Refusal of participation

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2021-05-03 (Actual); Primary Completion 2023-12-12 (Actual); Study Completion 2023-12-12 (Actual)

PRIMARY OUTCOMES:
Change in Body temperature | Day 1 , Day 60 , Day 90
  body temperature will be assessed using the bodyCap temperature monitor that records body temperature for up to 48h. this will be assessed for 24h on the three different phase (i) period of maintenance of body weight (CON); ii) two visits during weight loss (WL); iii) two visits during a weight regain (WG).)

SECONDARY OUTCOMES:
Body fat mass | Day 1 , Day 60 , Day 90
  the percentage of body fat will be assessed using X-ray absorptiometry (DXA)
  . This will be assessed on the three different phase (i) period of maintenance of body weight (CON); ii) two visits during weight loss (WL); iii) two visits during a weight regain (WG).)
Body fat free mass | Day 1 , Day 60 , Day 90
  the percentage of body fat free will be assessed using X-ray absorptiometry (DXA)
  . This will be assessed on the three different phase (i) period of maintenance of body weight (CON); ii) two visits during weight loss (WL); iii) two visits during a weight regain (WG).)
Food reward | Day 1 , Day 60 , Day 90
  The participants will be asked to complete a validated computer-based procedure to measure food reward (Leeds Food Preference Questionnaire; LFPQ) (Finlayson, King et al. 2008). This will be assessed on the three different phase (i) period of maintenance of body weight (CON); ii) two visits during weight loss (WL); iii) two visits during a weight regain (WG).)
Basal Metabolic rate | Day 1 , Day 60 , Day 90
  the resting energy expenditure will be assessed at rest during 30 minutes using indirect calorimetry (COSMED Fitmate Pro)
Cortisol | Day 1 , Day 60 , Day 90
  Cortisol concentrations will be assessed in the fasting state using salivary sample.
Measure of insulin mlUI/L | Day 1 , Day 60 , Day 90
  Insulin concentrations will be assessed in the fasting state using blood sample.
Measure of glucose g/L | Day 1 , Day 60 , Day 90
  Glucose concentrations will be assessed in the fasting state using blood sample.
Measure of triglycerides g/L | Day 1 , Day 60 , Day 90
  triglycerides concentrations will be assessed in the fasting state using blood sample.
Measure of LDL g/L | Day 1 , Day 60 , Day 90
  LDL concentrations will be assessed in the fasting state using blood sample.
Measure of HDL g/L | Day 1 , Day 60 , Day 90
  HDL concentrations will be assessed in the fasting state using blood sample.
Measure of cholesterol g/L | Day 1 , Day 60 , Day 90
  cholesterol concentrations will be assessed in the fasting state using blood sample.
Psychological profile | Day 1 , Day 60 , Day 90
  The psychological profile of the athletes will be assessed using the Profile of Mood state questionnaire that is a self-reported short pain and paper questionnaire.
Muscle strength | Day 1 , Day 60 , Day 90
  the muscle strength (in watt) will be assessed during a forced isometric contraction on a biodex.

CONTACTS AND LOCATIONS:
Overall Officials: Martine Duclos, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- Chu Clermont Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Derived] Bagot S, Ramos I, Miles-Chan J, Dulloo A, Hackney A, Boirie Y, Duclos M, Thivel D, Isacco L. The type of sport, but not sex, impacts body composition and metabolic response to a complete weight loss-weight regain episode in weight cycling athletes: results from the WAVE study. Appl Physiol Nutr Metab. 2025 Jan 1;50:1-13. doi: 10.1139/apnm-2024-0376. PMID 39919268